CLINICAL TRIAL: NCT00184041
Title: Treatment Of Newly Diagnosed Adult Acute Lymphoblastic Leukemia With Intensified Post Remission Therapy Containing PEG-Asparaginase.
Brief Title: Intensified Post Remission Therapy Containing PEG-Asparaginase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9L-03-1
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Daunorubicin; Vincristine; Prednisone; Methotrexate; pegaspargase; Mercaptopurine; Cyclophosphamide; Cytarabine; Teniposide; Thioguanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intensified Post-Remission: MTX/LV/PEG-Asparaginase (Experimental): Daunorubicin 60 mg/m2 iv on days 1, 2, 3 Vincristine 1.4 mg/m2 iv on days 1, 8, 15, 22 Peg-Asparaginase 2000 U/m2 iv on day 15 Prednisone 60 mg/m2 mg po on days 1-28 MTX 12 mg IT on days 8 & 15
  Interventions: Drug: Daunorubicin, Vincristine, Prednisone, Methotrexate, PEG-Asparaginase, 6-Mercaptopurine, Cytoxan, Cytosine Arabinoside, VM-26 and 6-Thioguanine

INTERVENTIONS:
Drug: Daunorubicin, Vincristine, Prednisone, Methotrexate, PEG-Asparaginase, 6-Mercaptopurine, Cytoxan, Cytosine Arabinoside, VM-26 and 6-Thioguanine — Induction I/II, consolidation I/II/III/IV and Maintenance

SUMMARY:
This study is for patients with recently diagnosed blood cancer, called acute lymphoblastic leukemia (ALL). The standard treatment for this disease consists of many chemotherapy drugs that are given in different combinations in several steps. Each step of treatment is called a cycle. Patients will be treated with the chemotherapy drugs that are routinely used in ALL and which are given in multiple treatment cycles over several months. All the chemotherapy drugs that are used in this study have been approved by the Food and Drug Administration (FDA).

One of the drugs, which is typically given to patients with ALL, is called Asparaginase. It is given together with the other drugs throughout the different cycles of treatment. This drug can be derived from several sources. The standard source is called E. coli Asparaginase, which is associated with a risk of allergic reactions. This drug stays in the body for a very short period of time; therefore, it has to be injected daily for 9-14 days in a cycle of treatment.

In this study, a different form of Asparaginase will be used, called PEG-Asparaginase (also called Oncospar), which remains in the body for about two weeks, therefore, it can be given only once in a cycle of treatment and still maintains high blood levels of the drug. PEG-Asparaginase has recently been approved by the FDA to treat ALL. Most of the experience with the drug has been in children with ALL. In children it was found to be as safe as the standard form of Asparaginase and with less allergic reaction. It was also found to have the same effectiveness on ALL. The experience with this drug in adults has been more limited.

The purpose of the study is to find out what side effects occur in adults when PEG-Asparaginase is given with other chemotherapy drugs and to see what effect it has on the response to treatment of ALL. Another purpose is to find out if the allergic reactions are reduced with PEG-Asparaginase. In children there is some early information that PEG-Asparaginase produces fewer antibodies than E.coli Asparaginase. Therefore, another purpose of the study is to see how many adult patients who receive PEG-Asparaginase develop antibodies against the drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients with previously untreated ALL subtypes L1 and L2.
* Patients with de novo Philadelphia (Ph)+ ALL (i.e. excluding those that are after blastic of CML) are eligible. However they will be referred to allogeneic hematopoietic stem cell transplantation and will continue on the study until they are ready to undergo the transplantation. At that time they will discontinue the study. Patients who are unable to undergo allogeneic transplantation will continue on the study.
* Presence of 25% or more of lymphoblasts in the bone marrow by FAB criteria, confirmed by TdT positivity or by flow cytometry with standard ALL markers.
* Patients may have received prior steroids.
* Age: 18 - 55 years
* Signed Informed Consent

Exclusion Criteria:

* Patients with Burkitt's ALL (L3 subtype) or CML lymphoblastic crisis are not eligible (including CML patients who present with ALL blastic crisis).
* Psychological or emotional disorders which will make a valid informed consent impossible.
* Bilirubin >1.5 mg/dl, creatinine > 2.5 mg/dl
* Symptomatic congestive heart failure or unstable angina
* Pregnant or lactating females
* Known HIV positive status

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2004-07; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Assessment of pt developing anti-asparaginase antibody | assessed 3 times

SECONDARY OUTCOMES:
Response | By Bone Marrow assessment

CONTACTS AND LOCATIONS:
Overall Officials: Dan Douer, MD, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California, United States

REFERENCES:
- [Derived] Douer D, Aldoss I, Lunning MA, Burke PW, Ramezani L, Mark L, Vrona J, Park JH, Tallman MS, Avramis VI, Pullarkat V, Mohrbacher AM. Pharmacokinetics-based integration of multiple doses of intravenous pegaspargase in a pediatric regimen for adults with newly diagnosed acute lymphoblastic leukemia. J Clin Oncol. 2014 Mar 20;32(9):905-11. doi: 10.1200/JCO.2013.50.2708. Epub 2014 Feb 10. PMID 24516026